CLINICAL TRIAL: NCT02083900
Title: Use of Banana Leaf Dressing on Donor Site Wounds: A Prospective Randomized Control Study
Brief Title: Use of Banana Leaf Dressing on Donor Site Wounds
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of the Philippines (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NIH (TRB) 2005-002
Record Dates: First submitted 2014-02-24; First posted 2014-03-11 (Estimated); Last update posted 2020-04-24 (Actual); Status verified 2020-04

CONDITIONS: Burn
MeSH Terms: conditions — Burns | interventions — Bandages, Hydrocolloid

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Banana Leaf Dressing Group (Experimental): The Banana Leaf Dressing site will receive a single layer of banana leaf dressing
  Interventions: Device: Banana Leaf Dressing
- Hydrocolloid Dressing Arm (Active Comparator): The donor under Hydrocolloid dressing was covered with hydrocolloid (DuoDERM CGF).
  Interventions: Drug: Hydrocolloid Dressing (DuoDERM CGF)

INTERVENTIONS:
Device: Banana Leaf Dressing — Banana leaf dressing will be prepared by cutting the mid rib of the leaf cutting the leaf into standard size of 12 x 12 inches to facilitate packing. The leaves are rolled and packed in polypropelene bags and subject to gamma irradiation or packed in paper bags for autoclaving. The Banana Leaf Dressing site will receive a single layer of banana leaf without any topical antibiotic applied to the wound followed by a layer of dry gauze for absorption of exudates. The dressing is secured with cling wrap to maintain an occlusive environment. This is then covered by rolled gauze and elastic bandage.
  Arms: Banana Leaf Dressing Group
Drug: Hydrocolloid Dressing (DuoDERM CGF) — The donor under HCD was covered with hydrocolloid (DuoDERM CGF). The hydrocolloid dressing was cut to the size of the donor site with an overlap of at least 2 centimeter around the wound edge. After pulling off the adhesive backing, care was taken to ensure that the adhesive was in direct contact with the raw surface. This was likewise covered with a top dressing of gauze for absorption of exudates and an elastic bandage to secure dressing.
  Other Names: DuoDERM CGF
  Arms: Hydrocolloid Dressing Arm

SUMMARY:
Prospective Randomized double-blind controlled trial comparing the healing rate, infection rate, pain score, ease of care and scar formation of Banana leaf dressing versus hydrocolloid dressing.

DETAILED DESCRIPTION:
Prospective Randomized double-blind controlled trial comparing the healing rate, infection rate, pain score, ease of care and scar formation of Banana leaf dressing versus hydrocolloid dressing.

Adult patients with no uncontrolled medical condition admitted at Philippine General Hospital Burn Center requiring split thickness skin graft for their burn. this is to compare the efficacy and safety of Banana Leaf Dressing with Hydrocolloid dressing among patients undergoing split thickness skin graft for their burn.

ELIGIBILITY:
Inclusion Criteria:

* Patient undergoing harvesting of skin graft one or both thigh
* Surgery under general anesthesia
* Given informed consent and has accomplished a written inform consent

Exclusion Criteria:

* Patient with uncontrolled medical condition such as diabetes or hypertension
* Pregnant females
* Patients in whom legs or back was used as donor site
* Surgery under regional anesthesia
* Refused inclusion into the study
* Patients who had previous skin harvesting on the area of the study

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2006-10; Primary Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Healing Assessment and Efficacy of the dressing | 8th post harvest day
  After 8th post harvest day The degree of healing will be assessed. Direct inspection of the wound will be made by experienced burn surgeon. The degree of re-epithelialization will be graded as follow:
  No Re-epithelialization = zero (0); Less than 50% = one (1); More than 50% but not complete = Two (2), and Complete (90% or more) = Three (3). Complete Re-epithelialization is synonymous to healing on which 90% or more of the wound surface is re-epithelialized.

SECONDARY OUTCOMES:
Pain Scores | taken from 24hours, on the 48th and 72 hour post skin harvest
  This pain score shall be determined on each patient using a visual analog pain intensity scale the score is as follows: 0-1=no pain; 2-3= Mild pain; 4-5=Moderate pain; 7-8= Severe pain; 9-10=Worst possible.

CONTACTS AND LOCATIONS:
Overall Officials: Jeane Azarcon, MD, Principal Investigator — UP Manila
Locations (1):
- Philippine General Hospital - University of the Philippines Manila, Manila, National Capital Region, Philippines